CLINICAL TRIAL: NCT05145543
Title: Effect of Topically Administered Levobupivacaine- Fentanyl Versus Levobupivacaine- Dexamethasone Combination in the Control of Pain After Endoscopic Sinus Surgery: A Randomized Controlled Trial
Brief Title: Effect of Topically Administered Levobupivacaine- Fentanyl Versus Levobupivacaine- Dexamethasone Combination in the Control of Pain After Endoscopic Sinus Surgery
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 17300428
Record Dates: First submitted 2021-11-26; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Endoscopic Sinus Surgery; Fentanyl
Keywords: dexamethasone; Levobupivacaine
MeSH Terms: interventions — Sodium Chloride; Levobupivacaine; Fentanyl; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group C (Placebo Comparator): 0.9 NaCl % (Saline) (5 ml)
  Interventions: Drug: Saline 0.9%
- Group L (Active Comparator): 0.25 % levobupivacaine (5 ml) will be applied.
  Interventions: Drug: Levobupivacaine Hydrochloride
- Group LF (Experimental): fentanyl plus 0.25 % levobupivacaine (5 ml) will be applied.
  Interventions: Drug: Levobupivacaine Hydrochloride; Drug: Fentanyl
- Group LD (Experimental): dexamethasone plus levobupivacaine (5 ml) will be applied.
  Interventions: Drug: Levobupivacaine Hydrochloride; Drug: Dexamethasone

INTERVENTIONS:
Drug: Saline 0.9% — 0.9 NaCl % (Saline) (5 ml) will be applied
  Arms: Group C
Drug: Levobupivacaine Hydrochloride — 0.25 % levobupivacaine (5 ml) will be applied.
  Arms: Group L; Group LD; Group LF
Drug: Fentanyl — fentanyl plus 0.25 % levobupivacaine (5 ml) will be applied.
  Arms: Group LF
Drug: Dexamethasone — Dexamethasone plus levobupivacaine (5 ml) will be applied.
  Arms: Group LD

SUMMARY:
Chronic sinusitis (CRS) is a high incidence disease characterized by pus, nasal obstruction, olfactory disturbance, headache, and other symptoms, lasting for more than 12 weeks, with severe cases having ocular compression and visual impairment, which can cause cranial, eye, and lung complications. Chronic sinusitis is a high-risk disease.

DETAILED DESCRIPTION:
One of the main concerns about using packing is that the removal is usually very painful and can be very bothersome. This procedure may even result in syncope by the activation of the vasovagal reflex system. There have been a few studies suggesting that nasal packs should not be used because removal from the nose causes serious discomfort and is painful. Many patients who have undergone nasal surgery report that the removal of the pack was the most painful part of the experience.

Postoperative pain is an acute inflammatory pain that starts with surgical trauma and ends with tissue healing. It can be harmful to organ systems by initiating inflamma¬tion through different mechanisms, and the alleviation of postoperative pain is considered important for obtaining homeostasis. Pain may initiate atelectasis due to improper coughing, immobilization may cause thromboembolism and catecholamine discharge may induce cardiovascular side effects and undesired changes in neuroendocrine or meta¬bolic function

ELIGIBILITY:
Inclusion Criteria:

* • ASA physical status I-II patients
* scheduled for elective FESS surgery. • Age from 18 to 65 years patients

Exclusion Criteria:

* • Age>18 and<65 years patients,

  * Previous history of FESS,
  * Patients with sensitivity to anesthetic agents in the study,
  * Patients who will do additional septoplasty or turbinate surgery,
  * Patients with disturbance of blood coagulation, including pro¬thrombin time (PT)/partial thromboplastin time (PTT) prolon¬gation, purpura, and spontaneous bleeding;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
time to first post-operative analgesic request | 24 hours postoperative
  when patient require analgesia

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut governorate, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Krings JG, Kallogjeri D, Wineland A, Nepple KG, Piccirillo JF, Getz AE. Complications of primary and revision functional endoscopic sinus surgery for chronic rhinosinusitis. Laryngoscope. 2014 Apr;124(4):838-45. doi: 10.1002/lary.24401. Epub 2013 Oct 9. PMID 24122737
- [Background] Chaaban MR, Rana N, Baillargeon J, Baillargeon G, Resto V, Kuo YF. Outcomes and Complications of Balloon and Conventional Functional Endoscopic Sinus Surgery. Am J Rhinol Allergy. 2018 Sep;32(5):388-396. doi: 10.1177/1945892418782248. Epub 2018 Jun 27. PMID 29947260
- [Background] Stankiewicz JA, Lal D, Connor M, Welch K. Complications in endoscopic sinus surgery for chronic rhinosinusitis: a 25-year experience. Laryngoscope. 2011 Dec;121(12):2684-701. doi: 10.1002/lary.21446. Epub 2011 Nov 15. PMID 22086769